CLINICAL TRIAL: NCT01668069
Title: Is Zofran Superior to Pyridoxine at Reducing Nausea and Vomiting in Pregnancy
Brief Title: Ondansetron VS Doxylamine and Pyridoxine in Treating Nausea of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP#NMCSD.2011.0151
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Vomiting of Pregnancy
Keywords: nausea; vomiting; pregnancy; ondansetron; doxylamine; vitamin B6; pyridoxine
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Experimental): study drug
  Interventions: Drug: Ondansetron
- Doxylamine and Pyridoxine (vitamin B6) (No Intervention): other nausea treatment in use

INTERVENTIONS:
Drug: Ondansetron — Ondansetron 4mg and a placebo capsule to be taken orally every 8 hours for 5 days.
  Other Names: Zofran
  Arms: Ondansetron

SUMMARY:
Our purpose is to determine whether ondansetron, a commonly used antiemetic, is equivalent in efficacy to the combination of pyridoxine and doxylamine, the currently recommended first line therapy for nausea and vomiting in pregnancy by the American Congress of Obstetricians and Gynecologists (ACOG). Since both treatments are safe in pregnancy, many physicians are using ondansetron as first line in practice. Despite this practice and the recommendations from ACOG, there is not data to suggest that ether practice is superior. This will be the first prospective, randomized, double blind, controlled trial comparing the two treatments. We hypothesize that ondansetron will be equally efficacious in reducing nausea and episodes of emesis. By alleviating nausea and vomiting associated with pregnancy, patients will likely benefit from less Emergency Department visits, urgent clinic visits, and admissions for progression to hyperemesis gravidarum.

ELIGIBILITY:
Inclusion Criteria:

* Women who are less than 16 weeks pregnant by last menstrual period or ultrasound
* Greater than 18 years of age
* English speaking
* No significant visual or hearing impairment
* Requesting treatment for nausea associated with pregnancy

Exclusion Criteria:

* If nausea or vomiting preexisted the pregnancy
* Requires hospitalization at the time of initial enrollment
* Already taking anti-emetics to include metoclopramide, ondansetron, doxylamine, pyridoxine, or promethazine
* The patient has an allergy to either study regimen
* If they are unable to return for a follow up visit in 1 week

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduction of nausea on the VAS (Visual Analog Scale) | 5 days

SECONDARY OUTCOMES:
Reduction in vomiting on the VAS | 5 days
Any adverse effects caused by the study medications. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Lauren G Oliveira, DO, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira LG, Capp SM, You WB, Riffenburgh RH, Carstairs SD. Ondansetron compared with doxylamine and pyridoxine for treatment of nausea in pregnancy: a randomized controlled trial. Obstet Gynecol. 2014 Oct;124(4):735-742. doi: 10.1097/AOG.0000000000000479. PMID 25198265